CLINICAL TRIAL: NCT04132895
Title: ICONIC: Improving Outcomes Through Collaboration in OsteosarComa
Acronym: ICONIC
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Bone Cancer Research Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: UCL/18/0248
Record Dates: First submitted 2019-07-02; First posted 2019-10-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Biobank; Genomics; Tumour markers; ImmuneOncology
MeSH Terms: conditions — Osteosarcoma | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin Fixed Paraffin Embedded (FFPE) archival blocks of tumour tissue removed during routine biopsy or surgery; Whole Blood Samples; New biopsies (FFPE & fresh frozen) obtained at relapse, or on resection of local recurrence/metastases.
  samples are optional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational only, no interventions are prescribed in protocol. — * Treatment will be given as per usual standard of care.
  * No treatments are specified by this protocol.

SUMMARY:
There has been little improvement in outcome for patients with osteosarcoma (OS) over the last 20 years. There have been only a few clinical trials of new treatments and no major new therapies introduced recently. This is in part because there is no good understanding of the biology of osteosarcoma, but also trials have only included subgroups of patients. The more that is understood about how and why osteosarcoma arises and grows the better clinicians will be able to decide what treatments are most likely to work best.

The purpose of this project is to collect high quality clinical data about patients of all ages with osteosarcoma, such as information about the size of the disease, how it was diagnosed and where it is at diagnosis, what treatments were given and how the disease responded the treatments.

Blood and tissue samples will also be collected for analysis in research laboratories. By looking at the results of the laboratory findings and the clinical data together, the questions will start to be answered about why osteosarcomas arise and grow, what makes it spread, and why some patients respond to treatment better than others. As time goes on, this information is planned to be used to develop clinical trials of new treatments.

Alongside this, the aim is to find out more about how osteosarcoma and its treatments affect the lives of those living with this disease. This information will help provide the most appropriate care and support that will meet the needs of each patient.

Ultimately, the aim is to improve the care and treatment of osteosarcoma patients so that they may live longer and better lives.

DETAILED DESCRIPTION:
Osteosarcoma is the most common bone sarcoma, accounting for approximately 30% of all bone sarcoma diagnoses. In England, it accounts for approximately 130 cases per year across all ages.

Generally osteosarcoma has an early peak in adolescent patients, with a second peak in patients over 60 years of age. There are differing treatments, including chemotherapy with more than one drug and surgery to the primary site - and for metastases where these occur.

Outcome, however, has improved little over the past 25 years with the proportion of patients surviving to 5 years remaining at about 42% for all ages and stages in the UK. Patients under 40 years of age (52%) are more likely to survive for 5 years than patients over 40 years (25%).

Survival also depends on the primary site of the osteosarcoma. It is poor for patients with tumours that are not in the limbs, at 36% for patients under the age of 40 years and as low as 6% for patients over 40 years. Also patients with metastatic disease at diagnosis still have a poor outcome.

The use of chemotherapy and surgery depends on factors such as age, the site of the osteosarcoma, how far spread it is and how well the patient is generally, with approximately two thirds of patients currently receiving chemotherapy, radiotherapy and surgery in England each year.

The most recent randomised trial for osteosarcoma, EURAMOS-1 [A randomized trial of the European and American Osteosarcoma Study Group to optimize treatment strategies for resectable osteosarcoma based on histological response to pre-operative chemotherapy], was an excellent example of an international effort to seek improved treatments for a rare cancer. Despite the participation of over 2000 patients, there were no changes to the standard of care for osteosarcoma.

There is still an unmet need to find new approaches, including biomarkers and new, targeted patient specific therapeutic approaches to improve outcomes for this group. This includes searching for improved systemic treatments and better approaches to management of the osteosarcoma. The ICONIC Study will provide a dataset for translational research into osteosarcoma.

Osteosarcoma clinical trials to date have focussed on a limited number of outcomes, usually in the younger patients with a tumour in a limb. So addressing complex inter-related questions has not been possible and several subpopulations of patients have not been studied. This limits opportunities to improve the standard of care. These groups include:

* patients with widely spread (metastatic) disease;
* patients with tumours in the less common locations such as the pelvis, spine and skull;
* patients with osteosarcoma with a background of skeletal abnormalities or an underlying genetic predisposition;
* the 50% of osteosarcoma arising in patients over 40 years.

Little is currently known about factors influencing treatment decisions in these groups and how consistently a standard of care is applied. The effect of treatments on quality of life, patient reported outcomes and other performance assessments is also not well described or understood. As osteosarcoma is quite rare it can be difficult for General Practitioners (GPs) to identify symptoms and patients often wait a long time before tests for osteosarcoma are carried out. How this affects outcomes is not known.

Overall, there is a need to broaden the ambition and scope of osteosarcoma research while improving access for all patients.

ELIGIBILITY:
Inclusion Criteria:

* New histological diagnosis of osteosarcoma or in the absence of osteoid seen on biopsy, pathology and imaging supportive of a diagnosis of osteosarcoma. (It is well recognised that some patients may present with features suggestive of osteosarcoma (under 40 years, radiological abnormality compatible) but in whom no osteoid is detected in needle biopsy. Although categorised as spindle cell tumour of bone, such patients are usually treated in an identical approach to osteosarcoma. A definite diagnosis of osteosarcoma is then often possible after surgery when the entire resection specimen is available.)
* Written informed consent of patient and/or parent/legal guardian.

Exclusion Criteria:

• Diagnosis more than four months prior to registration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with osteosarcoma in the UK at the time of the Study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility phase: Patient recruitment. | One year from study opening.
  To establish if a full study can be run, with a recruitment rate of ≥ 5 patients per month when 15 sites are open
Main Study: Patient recruitment | 3 years from study opening.
  Enrolment of at least 300 patients with blood and specimen samples at specified time points.

SECONDARY OUTCOMES:
Correlation of chemotherapy and radiotherapy to outcome | 4 years from registration.
  Correlation of chemotherapy and radiotherapy to outcome.
Do tumour margin and response to chemotherapy predict local recurrence in OS? | 4 years from registration.
  To use longitudinal data collected in the trial to predict local recurrence.
Correlation of tumour heterogeneity and clonal evolution to chemotherapy response and patient outcome. | 4 years from registration.
  Use of oncogenomic data collected in the trial to identify potential stratification for various regimens.
Validation of whole genome sequencing | 4 years from registration.
  Correlation of results from FFPE samples with whole genome sequencing results to identify potential stratification for various regimens.
Analysis of circulating biomarkers | 4 years from registration.
  Identification of potential tumour biomarkers for Osteosarcoma to predict burden of disease, response to therapy and outcome.
Patient reported outcomes | 4 years from registration.
  Assessment of the validity of the Sarcoma Assessment Measure (SAM) in osteosarcoma patients.
Analysis of PMBCs for IO research | 4 years from registration.
  Collection of Peripheral blood mononuclear cells in a cohort of patients for IO research

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Strauss, MD, Principal Investigator — University College Hospitals London
Locations (22):
- United Kingdom (22):
  - University College Hospitals London NHS Foundation Trust, London, Greater London
  - NHS Grampian Health Board, Aberdeen
  - Birmingham Women's and Childrens NHS Foundation Trust, Birmingham
  - The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University LHB, Cardiff
  - NHS Lothian Health Board, Edinburgh
  - NHS Greater Glasgow and Clyde Health Board, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Manchester University NHS Foundation Trust, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No